CLINICAL TRIAL: NCT03359512
Title: Comparison of Two Electroencephalograms (EEG) Monitors in Patients Undergoing General Anesthesia With Sevoflurane
Acronym: Bis-qCon-Hal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016/30; 2016-A01088-43 (Other: ANSM)
Record Dates: First submitted 2017-11-06; First posted 2017-12-02 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2017-11

CONDITIONS: General Anesthesia
Keywords: anesthesia monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- qCON monitor (Experimental): Simultaneous measurement of BIS and qCON
  Interventions: Device: qCON monitor

INTERVENTIONS:
Device: qCON monitor — supervision by qCON monitor of the depth of anesthesia

SUMMARY:
Quantium Medical Company has an ElectoEcenphalograph-based (EEG-based) algorithm with two outputs: qCON for unconsciousness and qNOX for anti-nociception. qCON, is designed to provide information about the depth of the hypnotic state, similar to that provided by the BIS™.

ELIGIBILITY:
Inclusion Criteria:

* Patients affiliated to a national insurance scheme or benefiting from such a program
* Patients having given their written consent.
* Patients that must benefit from a general anesthesia with the aim of a surgical act of a duration of at least one hour
* Patients that must benefit from a general anesthesia including a maintenance by the sevoflurane.
* For the patients taken care in ambulatory surgery, having a telephone and agreeing to communicate their phone number

Exclusion Criteria:

* Pregnant or breast-feeding Women
* Patients having a limit of use of the Bispectral Index (BIS) or qCON monitor ,
* Patients having a contraindication in the propofol.
* Patients taken care in ambulatory surgery who could not be contacted within 24 hours following the surgical operation;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-16 (Actual)

PRIMARY OUTCOMES:
qCON monitoring during maintenance of anesthesia | up to 10 hours
  Measurement of qCON values

SECONDARY OUTCOMES:
BIS monitoring during maintenance of anesthesia | One day
  Measurement of BIS values each 5 seconds during maintenance of anesthesia
qCON monitoring during induction of anesthesia | One day
  Measurement of qCON values each 5 seconds during induction of anesthesia
BIS monitoring during induction of anesthesia | One day
  Measurement of BIS values each 5 seconds during induction of anesthesia
qCON monitoring during recovery of anesthesia | One day
  Measurement of qCON values each 5 seconds during recovery of anesthesia
BIS monitoring during recovery of anesthesia during recovery of anesthesia | One day
  Measurement of BIS values each 5 seconds
Burst Suppression ratio retrieved by qCON monitoring | One day
  Measurement of Burst Suppression ratio values each 5 seconds during anesthesia
Burst Suppression ratio retrieved by BIS monitoring | One day
  Measurement of Burst Suppression ratio values each 5 seconds during anesthesia
qNOX monitoring during anesthesia | One day
  Measurement of qNOX values each 5 seconds during anesthesia
Periods of loss of signal of qCON | One day
  Measurement of qCON values each 5 seconds during anesthesia
Periods of loss of signal of BIS during anesthesia | One day
  Measurement of BIS values each 5 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Faiz Sofian, MD, Principal Investigator — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No